CLINICAL TRIAL: NCT06982261
Title: Voice2Manage: Interactive Voice-Assisted Self-Management Intervention for Low-Income Older Adults
Brief Title: Voice Technology-Based Self-Management Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Principal Investigator, Jane Chung, Acting Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00009631
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Low income older adults; Artificial Intelligence; Voice activated smart speakers (SS)
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Voice-activated smart speakers (Experimental): Participants will complete a set of standardized questionnaires. A list of smart speaker-based tasks will be introduced. Participants will then be asked to choose three tasks from a list.
  Interventions: Other: Voice-activated smart speakers

INTERVENTIONS:
Other: Voice-activated smart speakers — Participants will attend a single 90 to 120-minute in-person baseline visit to complete standardized questionnaires and review a list of smart speaker-based tasks. They will select three tasks; all will receive an Echo Show and a Fitbit Versa. Additional digital health devices (e.g., blood pressure monitor, in-home motion sensors) will be provided based on their selections. Participants will learn to interact with Alexa, followed by a second home visit one week later for task-specific setup and device installation.
  The team will conduct weekly or bi-weekly check-in calls for two months, with additional home visits as needed. At two months, a home visit will include questionnaires and a 30-60 minute interview on intervention feasibility. Participants will then use the devices independently for one month, with a final home visit at three months for questionnaires and a closing interview.

SUMMARY:
This study aims to test a new technology-based program designed to help improve the ability to manage chronic conditions.

This program includes daily smart speaker use for managing different tasks and technology learning.

Proper self-management of chronic conditions is critical to the maintenance of health. Digital technologies offer substantial potential to enhance self-management behaviors. Voice-operated smart speakers hold promise due to their ability to provide functional, cognitive, and social stimulation, send targeted reminders, and assist with daily schedules. Unfortunately, many older adults who live in low-income communities lack the resources and proficiency to take advantage of these options. Additionally, cognitive impairment is prevalent in independent living older adults, more prevalent in low-income older adults.

The goal is to address these critical challenges by identifying smart speaker-based functions preferred by older adults, exploring their technology challenges, introducing them to these functions, and providing necessary technology training to improve self-efficacy in managing chronic conditions and enhance their engagement in self-management behaviors.

DETAILED DESCRIPTION:
Many older adults live with two or more chronic diseases. These conditions impact functional impairment and quality of life. Inadequate management of chronic conditions significantly burdens individuals and society, accounting for 75% to 90% of total healthcare expenditures in the United States. Proper self-management, the ability to manage symptoms, treatments, lifestyle changes, and psychosocial, cultural, and spiritual consequences of chronic conditions, is critical to effective chronic disease management. Central to this successful self-management is the concept of self-efficacy, a person's belief in their ability to accomplish specific tasks or particular goals. Digital technologies offer substantial potential to enhance self-management of chronic conditions. Unfortunately, many older adults living on a low income lack the resources and proficiency to take advantage of these options. Additionally, cognitive impairment is prevalent in independent-living older adults, which affects the ability to manage everyday health needs.

Voice-activated smart speakers (SS; e.g., Amazon Echo) especially hold promise due to their ability to provide functional, cognitive, and social stimulation, send targeted reminders, and assist with daily schedules. However, these devices and their applications are not always intuitive. Our preliminary studies demonstrated critical challenges in SS adoption and use in low-income older adults, such as difficulty setting up key SS functions or finding relevant resources or information necessary for figuring out the process. The challenges arose from various factors, including insufficient training and technical support, low health literacy, and cognitive impairments. Crucial to the successful use of SS to support low-income older adults, some initial development stages are necessary.

Researchers' overall objective in this research is to test the feasibility, acceptability, and preliminary efficacy of an interactive SS-based self-management intervention for low-income older adults living with chronic conditions and mild cognitive impairment. The study team will first identify SS functions preferred by this group of older adults and strategies to support their learning of SS-based functions for self-management of chronic conditions, and deploy them in older adults' homes to manage chronic conditions

ELIGIBILITY:
Inclusion Criteria:

* Persons 55 years of age and older,
* Living in subsidized housing or with a housing voucher and having an annual income less than $30K,
* One or more chronic conditions,
* Having probable mild cognitive impairment (MCI), based on the education-adjusted Montreal Cognitive Assessment (MoCA) score less than 24 and greater than or equal to 18,
* Living alone independently, and
* Able to speak and read English.

Exclusion Criteria:

* Severe visual/hearing impairment requiring assistance in participating in interactions with the smart speaker and integrated devices,
* Self-reported diagnoses of Alzheimer's disease and related dementias,
* Significant medical illness interfering with the study assessments and activities,
* Inability to provide informed consent, and
* Nursing home residents.
* Eligibility will not be limited to smart speaker ownership.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Retention Rate | 3 months
  Retention rate will be measured by the number of individuals who continue participating in a program for up 3 months
System Usability Scale | Baseline, 2 months, and 3 months
  Acceptance will be measured using the System Usability Scale (SUS) that is a widely used, validated tool for measuring the perceived usability of a system (e.g., software, website, device). It consists of 10 items, each rated on a 5-point Likert scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree). The researcher will modify the wording slightly to make the questions appropriate for the technology system being evaluated.
  Score > 68: Above average usability Score = 68: Average usability benchmark Score < 68: Below average usability
Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v1.0 Self-Efficacy for Managing Chronic Conditions - Managing Medications and Treatment | Baseline, 2 months, and 3 months
  The PROMIS Item Bank v1.0 Self-Efficacy measure assesses self-reported current level of confidence in managing chronic conditions, with a focus on managing medications and treatment regimen related to chronic health conditions. It consists of 26 items, each rated on a 5-point Likert scale ranging from 1 (not at all confident) to 5 (very confident). Raw scores (sum of item responses) are converted to T-scores using the PROMIS scoring system. A score of 50 is the average for the United States general population, with a standard deviation of 10. Higher T-scores indicate greater self-efficacy in managing medications and treatment.
Self-Care of Chronic Illness Inventory (V.4C) | Baseline, 2 months, and 3 months
  The Self-Care of Chronic Illness Inventory (SC-CII) version 4c is a validated tool designed to assess self-care behaviors in individuals managing chronic illnesses. Each item within the SC-CII is rated on a 5-point Likert scale, typically ranging from 1 ("Never") to 5 ("Always"). It evaluates self-care across three key domains: Self-Care Maintenance (Section A), Self-Care Monitoring (Section B), and Self-Care Management (Section C). Also, it examines Self-Care Confidence (Section D).
  Scores for each domain are calculated by summing the item responses within that domain. Higher scores indicate better self-care behaviors in the respective domain. A standardized score of 70 or above in any domain is generally considered indicative of adequate self-care. Scores below 70 may suggest areas where the individual could benefit from additional support or intervention to enhance self-care practices.
Modified Computer Self-Efficacy Scale | Baseline, 2 months, and 3 months
  Modified Computer Self-Efficacy Scale (mCSES) is a modification of Compeau and Higgins 10-item Computer Self-Efficacy Scale, developed to make it applicable for clinical settings (for use with older people or people with disabilities using everyday technologies). The questions ask to indicate whether "you could use this unfamiliar technology under a variety of conditions". Rated on a 10-point scale of confidence. Principal components analysis yields a two-factor structure: 1. Using the Technology Alone (e.g., "If there was no one around to tell me what to do as I go"), and 2. Using the Technology with the Support of Others (e.g., " If someone else had helped me get started"). Participants with higher levels of technology self-efficacy would be more frequent users of everyday technology.
Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Adult Profile questionnaire | Baseline, 2 months, and 3 months
  The PROMIS-29 Adult Profile measure assesses pain intensity using a single 0-10 numeric pain rating item and seven health domains using four items each: physical functioning, fatigue, pain interference, depression, anxiety, ability to participate in social roles and activities, and sleep disturbance. Each item is rated on a Likert-type scale, typically 1 (not at all) to 5 (very much), with response options indicating the frequency or severity of symptoms or experiences. For most PROMIS instruments, a score of 50 is the average for the United States general population, with a standard deviation of 10. Higher scores for Depression, Fatigue, Sleep Disturbance, and Pain Interference indicate worse health than average.
Engagement in Self-Management Behaviors determined by smart speaker interaction logs | 2 months and 3 months
  The research team will extract the text-based Alexa usage data showing verbal commands used by each participant to examine types of verbal commands, frequency, and regularity of smart speaker use to determine participants' engagement in self-management behaviors.

SECONDARY OUTCOMES:
Factors affecting the implementation and dissemination of the Voice2Manage | 2 months and 3 months
  Open ended questions to assess possible factors affecting implementation and dissemination. No scoring scale is available.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Chung, PhD, RN, Principal Investigator — Emory University - Nell Hodgson Woodruff School of Nursing
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available to qualified researchers.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after publication.
Access Criteria: Requests will be reviewed by the study's PI. Approved requesters will receive data through a secure data transfer platform following execution of a data use agreement.